CLINICAL TRIAL: NCT04262505
Title: A MEDiterranean Diet in Rheumatoid Arthritis (MEDRA)
Brief Title: A MEDiterranean Diet in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, Tala Raad, PhD Candidate, University of Limerick
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDRA
Record Dates: First submitted 2020-02-04; First posted 2020-02-10 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Mediterranean diet; Randomised controlled trial; Ireland
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Mediterranean diet vs. Irish healthy eating guidelines
Masking Description: Due to the nature of dietary interventions, blinding will not be possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet Group (Group A) (Experimental): The intervention is based on components of the traditional Mediterranean diet which is primarily a plant based diet and emphasises intakes of vegetables, whole grains and fruit with the main added fat being extra virgin olive oil.The diet will be modified and tailored to cultured preferences by the registered dietitian. Participants will be informed of their diet allocation group during the baseline teleconsultation and will commence the diet the following day or as soon as is feasible for 12 weeks. Participants will be provided with resources specifically designed to explain the components of the Mediterranean diet and how it will be followed.
  Interventions: Behavioral: Mediterranean Diet Group
- Healthy Eating Group (Group B) (Experimental): Participants assigned to the Healthy Eating group will be advised to adhere to the current healthy eating guidelines and will be provided with resources to inform them of these guidelines and sample meal plans that are readily available on the Healthy Ireland website.
  Interventions: Behavioral: Healthy Eating Group

INTERVENTIONS:
Behavioral: Mediterranean Diet Group — Participants will be advised to follow a traditional Mediterranean diet
  Arms: Mediterranean Diet Group (Group A)
Behavioral: Healthy Eating Group — Participants will be advised to follow the Healthy Eating Guidelines in Ireland
  Arms: Healthy Eating Group (Group B)

SUMMARY:
The MEDRA study is a 12-week randomised controlled trial that aims to assess effects of a Mediterranean dietary telehealth intervention compared to the Irish Healthy Eating guidelines on the physical function and quality of life of adults living with Rheumatoid Arthritis in Ireland. Investigators will be able to determine how closely people living in Ireland can accept the Mediterranean dietary practices and adhere to them with dietetic input and guidance.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a long-term inflammatory disease which commonly occurs in the small joints of the hands, wrists and feet leading to swelling, pain and stiffness in the affected joints. The condition is two to three times more prevalent in women than in men. Although it might occur at any age, the incidence of the disease is highest between the ages of 40 and 65 years. Currently, there is no treatment that provides complete remission of the disease for people living with RA. Treatment of RA aims to reduce the symptoms and improve the health of the patient. Although diet is not part of the mainstream treatment, many studies have reported beneficial effects of certain diets on RA symptoms. The MEDRA study will examine the habitual dietary intakes of people living with RA in Ireland and will explore whether people with RA will benefit from either a Mediterranean dietary pattern or the Healthy eating guidelines in Ireland. This small scale study will provide useful information on whether people with RA in Ireland can adhere to a Mediterranean dietary pattern and whether the intervention will have beneficial impact on the physical function and quality of life. This is important work prior to proceeding to larger intervention studies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year
* Definite diagnosis of rheumatoid arthritis according to ACR or EULAR criteria
* Full access to Internet/smartphone
* English speaking

Exclusion Criteria:

* Age <18 years
* Breastfeeding, pregnant or trying to get pregnant.
* Patients who have commenced nutritional supplements or a new dietary regime in the month prior to study enrolment.
* Patients who do not have access to the Internet/smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Changes in Quality of Life | Throughout the 12 weeks study period (At baseline, mid-intervention and post-intervention)
  Rheumatoid Arthritis Quality of Life questionnaire (RAQoL) will be used to describe the individuals' perceptions, satisfaction, and evaluation of different areas of their own lives, such as physical health and functioning, psychological and emotional well-being, social roles, and relationships. A scale 1 to 30 will be used whereby the higher the score, the worse the QoL.
Changes in Physical Function | Throughout the 12 weeks study period (At baseline, mid-intervention and post-intervention)
  The health assessment questionnaire disability index (HAQ-DI) is an index used to assess how arthritis impacts the participant's everyday life. A scale 0-3 is used whereby 3 indicated very severe disability.

SECONDARY OUTCOMES:
Change in Diet adherence | Throughout the 12 weeks study period (At baseline, mid-intervention and post-intervention)
  Assessment of participants' adherence to either the Mediterranean diet or the current Irish Healthy Guidelines will be assessed using a PREDIMED validated checklist and a Healthy Eating checklist respectively. Higher scores indicate greater adherence to the diet assigned. A 3-day food diary will also be used to captures the dietary intake of participants
Change in Physical activity levels | Throughout the 12 week study period (At baseline, mid-intervention and post-intervention)
  Assessment of participants' physical activity levels using the YPAS (Yale Physical activity survey)

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Tierney, Principal Investigator — Unievrsity of Limerick
Locations (1):
- University Hospital Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Raad T, George E, Griffin A, Larkin L, Fraser A, Kennedy N, Tierney A. Effects of a telehealth-delivered Mediterranean diet intervention in adults with Rheumatoid Arthritis (MEDRA): a randomised controlled trial. BMC Musculoskelet Disord. 2024 Aug 7;25(1):631. doi: 10.1186/s12891-024-07742-1. PMID 39112976
- [Derived] Raad T, George E, Griffin A, Larkin L, Fraser A, Kennedy N, Tierney A. A randomised controlled trial of a Mediterranean Dietary Intervention for Adults with Rheumatoid Arthritis (MEDRA): Study protocol. Contemp Clin Trials Commun. 2022 May 3;28:100919. doi: 10.1016/j.conctc.2022.100919. eCollection 2022 Aug. PMID 35620325